CLINICAL TRIAL: NCT06187805
Title: Retrospective Case Series Evaluating the Outcome of Transcrestal Sinus Elevation Using Autogenous Bone Supporting an OSSIX Volumax Collagen Xenograft Scaffolding
Brief Title: Retrospective Case Series - OSSIX Volumax Collagen Xenograft Scaffolding
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Old Orchard Periodontics and Implant Dentistry LTD (Other)
Responsible Party: Sponsor
Other Study IDs: Ver 01
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Dental Implants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Up to 15 patients: Patients who have had a transcrestal elevation using autogenous bone supporting an OSSIX Volumax collagen scaffolding.
  Interventions: Device: OSSIX Volumax

INTERVENTIONS:
Device: OSSIX Volumax — OSSIX Volumax is used in combination with autogenous bone collected during preparation of the implant osteotomy.

SUMMARY:
This study is designed as a retrospective, single center study. Up to 15 participants who had a transcrestal sinus elevation and implant placement using autogenous bone supporting an OSSIX Volumax collagen xenograft scaffolding will be enrolled. The study will include data collection from medical records and data collected at a follow up visit between January 2019 and March 2023.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the outcome of transcrestal sinus elevation using autogenous bone supporting an OSSIX Volumax collagen scaffolding. Data to be collected includes demographics, past medical history including autoimmune diseases and connective tissue diseases, smoking history and known allergies. Implant data will be collected and change in crestal bone height will be measured radiographically and cone beam computed tomography at follow up. The protocol will include both single-staged and two-staged procedures. Adverse events will be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

1. Transcrestal sinus lift planned
2. Implant therapy planned
3. Crestal bone height < or equal to 6mm
4. Missing tooth or teeth for function
5. Nonsmoker -

Exclusion Criteria:

1. Patients with known collagen hypersensitivity
2. Patients with sensitivity to porcine-derived materials
3. Patients suffering from autoimmune diseases and connective tissue diseases, such as lupus erythematosus, dermatomyositis, etc.
4. Pregnant or planning to become pregnant (verbal confirmation)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 15 participants who meet the I/E will have data retrospectively reviewed and will include follow up data.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in crestal bone height | 4 months to 57 months
  Measured radiographically and by cone beam computed tomography at follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Old Orchard Periodontics and Implant Dentistry, Skokie, Illinois, United States